CLINICAL TRIAL: NCT03870854
Title: Paced Electrogram Feature Analysis (PEFA) for Ablation Targeting in Ischaemic Ventricular Tachycardia
Acronym: PEFA-VT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Damian Redfearn (Other)
Responsible Party: Sponsor-Investigator, Dr. Damian Redfearn, MB CHB MD MRCPI FRCPC Professor of Medicine, Kingston Health Sciences Centre, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-PA #1723
Record Dates: First submitted 2019-03-06; First posted 2019-03-12 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Ventricular Tachycardia (VT)

STUDY DESIGN:
Intervention Model Description: This is a Canadian multi-centre prospective cohort study of 40 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEFA targeted substrate ablation (Experimental): Use of PEFA strategy to identify and target VT isthmuses.
  Interventions: Procedure: PEFA VT ablation technique

INTERVENTIONS:
Procedure: PEFA VT ablation technique — Catheter ablation guided by PEFA technique
  Other Names: Paced electrogram feature analysis or 'PEFA'

SUMMARY:
Canadian multicentre prospective cohort study of 40 patients with ischaemic heart disease and therapy from an implantable cardioverter defibrillator (ICD).

DETAILED DESCRIPTION:
Paced Electrogram Feature Analysis is employed to elucidate VT isthmus sites and target Type I sites for ablation to prevent recurrent VT/VF.

The trial hypothesis is: catheter ablation employing PEFA will, in comparison to published data, reduce the composite outcome of death at any time, appropriate ICD shock, ventricular tachycardia storm or treated sustained ventricular tachycardia below the detection rate of the ICD or incessant VT for patients with prior myocardial infarction and sustained ventricular tachycardia or fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years of age
* Ischaemic heart disease and prior myocardial infarction (using the international definition of MI: Q waves or imaging evidence of regional myocardial akinesis/thinning in the absence of a non-ischemic cause with documentation of prior ischaemic injury)
* Eligible for catheter ablation as standard of care
* Implantable Cardioverter Defibrillator

Exclusion Criteria:

* Unable or unwilling to provide consent
* Both mechanical aortic and mitral valve
* LV thrombus,
* NYHA class IV heart failure symptoms
* Contraindication to heparin
* Survival limited to <1 year in estimation of attending care team,
* Prior VT ablation Exclusion to standard of care VT catheter ablation procedure such as
* Active ischaemia (acute thrombus diagnosed by coronary angiography, or dynamic ST segment changes demonstrated on ECG) or another reversible cause of VT (e.g. drug- induced arrhythmia), had recent acute coronary syndrome within 30 days thought to be due to acute coronary arterial thrombosis, or have CCS functional class IV angina. Note that biomarker level elevation alone after ventricular arrhythmias does not denote acute coronary syndrome or active ischemia.
* Non-ischaemic cardiomyopathy because of reduced ablation success and PEFA has not been examined in the context of a non-ischaemic cardiomyopathy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 3 years
  a composite of death - any time post procedure myocardial infarction and sustained ventricular tachycardia or fibrillation.
Appropriate ICD shock | 3 years
  Time to first appropriate ICD shock - any time post procedure
VT storm | 3 years
  Time to 3 or more episodes of VT within 24 hours - any time post procedure
Treated sustained VT below the detection rate of the ICD | 3 years
  Time to any sustained VT below the detection rate of the ICD; e.g. by external cardioversion, pharmacologic conversion, or manual ICD therapy - any time post procedure
Incessant VT | 3 years
  Time to incessant VT defined as a sustained ventricular arrhythmia which does not terminate despite appropriate external cardioversion/defibrillation or ICD antitachycardia pacing or shocks, or terminates but reinitiates within ≤5 seconds - any time post procedure

SECONDARY OUTCOMES:
Appropriate anti-tachycardia pacing (ATP) from ICD | 3 years
  Appropriate anti-tachycardia pacing (ATP) from ICD - any time post procedure
Inducible for ventricular arrhythmia | 3 years
  Number of inducible for ventricular arrhythmia following catheter ablation guided by PEFA protocol
Number of ventricular arrhythmia events | 3 years
  This is a composite of appropriate ATP, appropriate shock, sustained VT not treated by ICD, external cardioversion, or pharmacologic cardioversion, and incessant VT - any time during or after the procedure
Escalation and De-escalation of antiarrhythmic medication | 3 years
  Any increase or decrease in the dosage of antiarrhythmic medication either due to inefficacy or side effects will be assessed - any time post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Damian Redfearn, MD, Principal Investigator — Queen's University
Locations (3):
- Canada (3):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institutation, Ottawa, Ontario